CLINICAL TRIAL: NCT01667900
Title: Pharmacokinetics of a Single Dulaglutide Dose in Healthy Chinese Subjects and of Multiple Dulaglutide Doses in Chinese Patients With T2DM
Brief Title: A Study of Dulaglutide in Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12925; H9X-EW-GBDL (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 0.5 mg Dulaglutide (Part A-Healthy) (Experimental): 0.5 milligrams (mg) dulaglutide administered once subcutaneously (SQ) to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Dulaglutide; Drug: Placebo
- 0.75 mg Dulaglutide (Part A-Healthy) (Experimental): 0.75 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Dulaglutide; Drug: Placebo
- 1.5 mg Dulaglutide (Part A-Healthy) (Experimental): 1.5 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Dulaglutide; Drug: Placebo
- Placebo (Part A-Healthy) (Placebo Comparator): Placebo administered once SQ to healthy participants in 1 of 3 treatment periods
  Interventions: Drug: Placebo
- 0.5 mg Dulaglutide (Part B-T2DM) (Experimental): 0.5 mg dulaglutide administered to participants with Type 2 diabetes mellitus (T2DM) once weekly SQ for 4 weeks
  Interventions: Drug: Dulaglutide; Drug: Placebo
- 0.75 mg Dulaglutide (Part B-T2DM) (Experimental): 0.75 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks
  Interventions: Drug: Dulaglutide; Drug: Placebo
- 1.5 mg Dulaglutide (Part B-T2DM) (Experimental): 1.5 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks
  Interventions: Drug: Dulaglutide; Drug: Placebo
- Placebo (Part B-T2DM) (Placebo Comparator): Placebo administered to participants with T2DM once weekly SQ for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide
  Other Names: LY2189265
  Arms: 0.5 mg Dulaglutide (Part A-Healthy); 0.5 mg Dulaglutide (Part B-T2DM); 0.75 mg Dulaglutide (Part A-Healthy); 0.75 mg Dulaglutide (Part B-T2DM); 1.5 mg Dulaglutide (Part A-Healthy); 1.5 mg Dulaglutide (Part B-T2DM)
Drug: Placebo — Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.

SUMMARY:
This is a study of dulaglutide in Chinese participants. The purpose of the study is to determine how the body processes dulaglutide and how dulaglutide affects the body. This study has 2 parts: Part A - single dose of dulaglutide administered to healthy participants in 2 of 3 study periods. There is a minimum 28-day washout between periods. Part A will last approximately 16 weeks. Part B - multiple doses of dulaglutide administered to participants with Type 2 diabetes mellitus (T2DM). Part B will last approximately 15 weeks.

Doses of 0.5 milligrams (mg), 0.75 mg, and 1.5 mg of dulaglutide will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Native Chinese (all 4 grandparents of Chinese origin)
* Male participants with female partners of child-bearing potential, or partners who are pregnant or breastfeeding, agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator.
* The method of contraception may be one of the following: condom with spermicidal agent, male participant sterilization, true abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable).
* Female participants not of child-bearing potential (i.e. are postmenopausal or permanently sterilized [e.g. tubal occlusion, hysterectomy, bilateral salpingectomy]). Such participants will not be required to use contraception but must test negative for pregnancy at the time of enrollment. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) or at least 1 year of spontaneous amenorrhea, with follicle stimulating hormone (FSH) ≥40 milli international units per milliliter (mIU/mL).
* Female participants who have undergone sterilization by tubal ligation: agree to use a condom in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of investigational product. Such participants must also test negative for pregnancy at the time of enrollment.

Participants with T2DM:

* Have T2DM controlled with diet or exercise alone or with a single oral agent antihyperglycemic medication (OAM) (metformin, sulfonylureas, meglitinides, acarbose [or other disaccharidase inhibitors] or thiazolidinediones) for at least 3 weeks (3 months for thiazolidinediones) before admission. Note that participants receiving sulfonylureas, meglitinides or acarbose may participate only if this treatment is stopped and metformin substituted. If switched to metformin, participants should be allowed to stabilize on metformin for 3 weeks before receiving study drug.
* If T2DM controlled with diet or exercise alone, must have a hemoglobin A1c (HbA1c) value of 6.5% to 10.5% at screening and a fasting blood glucose value of 126 to 250 milligrams per deciliter (mg/dL) (approximately 7.0 to 13.9 millimoles per liter [mmol/L]) at screening.
* If T2DM controlled with OAM(s), must have an HbA1c value of 9.0% or less at screening and a fasting blood glucose value of 110 to 200 mg/dL (approximately 6.1 to 11.1 mmol/L) at screening. If a participant's T2DM is being controlled with OAM(s) other than metformin, the participant's OAM will be stopped for at least 3 weeks before administration of study drug.

Exclusion Criteria:

All Participants:

* Have a history or presence of cardiovascular (myocardial infarction, cerebrovascular accident, venous thromboembolism), respiratory, hepatic, renal, hematological, neurological autoimmune or endocrine (except T2DM), disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have evidence of significant active neuropsychiatric disease.
* Have poorly controlled hypertension (systolic >160 millimeters of mercury [mmHg] and/or diastolic >100 mmHg) and/or evidence of labile blood pressure including symptomatic postural hypotension.
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric empty (for example, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or dipeptidyl peptidase (DPP)-4 inhibitors. Participants with dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician.
* Have personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC.

Participants with T2DM

* Have experienced outpatient use of insulin for control of diabetes within the past 6 months.
* Have clinically significant peripheral vascular occlusive disease in the opinion of the investigator.
* Have known severe exudative diabetic retinopathy in the opinion of the investigator.
* Have known significant autonomic neuropathy as evidenced by urinary retention, diabetic diarrhea, or gastroparesis.
* Have experienced a ketoacidotic episode (pH less than 7.3) requiring hospitalization in the last 6 months.
* Regular use of drugs that affect the glycodynamics and that directly reduce gastrointestinal motility (eg, anticholinergics, antispasmodics, 5HT3 antagonists, dopamine antagonists, and opiates) and of systemic corticosteroids by oral, intravenous, or intramuscular route, or potent, inhaled, or intranasal steroids known to have a high rate of systemic absorption.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM- 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing, China

REFERENCES:
- [Derived] Xu J, Zhang Y, Li Y, Zhao X, Zhou W, Loghin C, Tham LS, Cui X, Cui Y, Wang W. Pharmacokinetics, Pharmacodynamics, and Safety of Dulaglutide After Single or Multiple Doses in Chinese Healthy Subjects and Patients with T2DM: A Randomized, Placebo-Controlled, Phase I Study. Adv Ther. 2022 Jan;39(1):488-503. doi: 10.1007/s12325-021-01921-5. Epub 2021 Nov 17. PMID 34787823

RESULTS

PARTICIPANT FLOW:
Groups:
- First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.5 milligrams (mg) dulaglutide administered once subcutaneously (SQ)
  Period 2: placebo administered once SQ
  Period 3: 1.5 mg dulaglutide administered once SQ
- First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.75 mg dulaglutide administered once SQ
  Period 2: 0.5 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.75 mg dulaglutide administered once SQ
  Period 2: 1.5 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.5 mg dulaglutide administered once SQ
  Period 2: 1.5 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 1.5 mg dulaglutide administered once SQ
  Period 2: placebo administered once SQ
  Period 3: 0.75 mg dulaglutide administered once SQ
- First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: placebo administered once SQ
  Period 2: 0.5 mg dulaglutide administered once SQ
  Period 3: 1.5 mg dulaglutide administered once SQ
- First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.75 mg dulaglutide administered once SQ
  Period 2: placebo administered once SQ
  Period 3: 1.5 mg dulaglutide administered once SQ
- First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: placebo administered once SQ
  Period 2: 0.75 mg dulaglutide administered once SQ
  Period 3: 0.5 mg dulaglutide administered once SQ
- First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: placebo administered once SQ
  Period 2: 0.75 mg dulaglutide administered once SQ
  Period 3: 1.5 mg dulaglutide administered once SQ
- First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.5 mg dulaglutide administered once SQ
  Period 2: 0.75 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 1.5 mg dulaglutide administered once SQ
  Period 2: 0.75 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.5 mg dulaglutide administered once SQ
  Period 2: placebo administered once SQ
  Period 3: 0.75 mg dulaglutide administered once SQ
- First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 0.75 mg dulaglutide administered once SQ
  Period 2: placebo administered once SQ
  Period 3: 0.5 mg dulaglutide administered once SQ
- First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: placebo administered once SQ
  Period 2: 1.5 mg dulaglutide administered once SQ
  Period 3: 0.75 mg dulaglutide administered once SQ
- First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: 1.5 mg dulaglutide administered once SQ
  Period 2: 0.5 mg dulaglutide administered once SQ
  Period 3: placebo administered once SQ
- First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy): Part A involved overtly healthy participants and was comprised of 3 treatment periods. There was a washout period of at least 28 days between doses.
  Period 1: placebo administered once SQ
  Period 2: 1.5 mg dulaglutide administered once SQ
  Period 3: 0.5 mg dulaglutide administered once SQ
- 0.5 mg Dulaglutide (Part B-T2DM): 0.5 mg dulaglutide administered to participants with Type 2 diabetes mellitus (T2DM) once weekly SQ for 4 weeks in Part B
- 0.75 mg Dulaglutide (Part B-T2DM): 0.75 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks in Part B
- 1.5 mg Dulaglutide (Part B-T2DM): 1.5 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks in Part B
- Placebo (Part B-T2DM): Placebo administered to participants with T2DM once weekly SQ for 4 weeks in Part B
Period: Part A, Period 1
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 (Part B participants did not participate in Part A.) | 0 (Part B participants did not participate in Part A.) | 0 (Part B participants did not participate in Part A.) | 0 (Part B participants did not participate in Part A.)
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Washout 1
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Period 2
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Washout 2
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A, Period 3
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | First 0.5 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First 0.75 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then 1.5 mg, Then Placebo (Part A-Healthy) | First 1.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First Placebo, Then 0.5 mg, Then 1.5 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 1.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 0.75 mg, Then 1.5 mg (Part A-Healthy) | First 0.5 mg, Then 0.75 mg, Then Placebo (Part A-Helathy) | First 1.5 mg, Then 0.75 mg, Then Placebo (Part A-Healthy) | First 0.5 mg, Then Placebo, Then 0.75 mg (Part A-Healthy) | First 0.75 mg, Then Placebo, Then 0.5 mg (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.75 mg (Part A-Healthy) | First 1.5 mg, Then 0.5 mg, Then Placebo (Part A-Healthy) | First Placebo, Then 1.5 mg, Then 0.5 mg (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM)
Started | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 0 (Part A participants did not participate in Part B.) | 11 | 11 | 10 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 11 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Part A-Healthy: Part A (single-dose, 3 treatment period, crossover design) involved overtly healthy participants only. Each participant received single doses of placebo and 2 of the 3 dulaglutide doses (0.5, 0.75, and 1.5 mg), in 3 treatment periods, such that placebo was administered SQ to all 16 participants and 0.5, 0.75, and 1.5 mg dulaglutide was administered SQ to 10, 11, and 11 participants, respectively. There was a washout period of at least 28 days between doses.
- 0.5 mg Dulaglutide (Part B-T2DM): 0.5 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks in Part B
- Total: Total of all reporting groups
Arm/Group | Part A-Healthy | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM) | Total
Number analyzed (Participants) | 16 | 11 | 11 | 10 | 10 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (5.6) | 58.2 (4.2) | 56.9 (13.1) | 55.8 (8.5) | 51.8 (8.3) | 48.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 3 | 3 | 12
  Male | 16 | 8 | 8 | 7 | 7 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 11 | 11 | 10 | 10 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 16 | 11 | 11 | 10 | 10 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 16 | 11 | 11 | 10 | 10 | 58

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Dulaglutide
Description: Pharmacokinetic parameters were assessed on Day 1 in Part A and Days 1 and 22 in Part B.
Time Frame: Pre-dose and 12, 24, 48, 72, 96, 168, and 336 hours post-dose
Population: Participants in Part A and Part B who received at least 1 dose of study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 0.5 mg Dulaglutide (Part A-Healthy): 0.5 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods in Part A
- 0.75 mg Dulaglutide (Part A-Healthy): 0.75 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods in Part A
- 1.5 mg Dulaglutide (Part A-Healthy): 1.5 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods in Part A
Arm/Group | 0.5 mg Dulaglutide (Part A-Healthy) | 0.75 mg Dulaglutide (Part A-Healthy) | 1.5 mg Dulaglutide (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM)
Number analyzed (Participants) | 10 | 11 | 11 | 11 | 11 | 10
nanograms per milliliter (ng/mL)
  Day 1 (Parts A and B) | 29.4 (39) | 44.2 (14) | 81.5 (21) | 20.7 (18) | 31.3 (23) | 52.6 (28)
  Day 22 (Part B only) | NA (NA) — Part A participants did not have data collected at this time point | NA (NA) — Part A participants did not have data collected at this time point | NA (NA) — Part A participants did not have data collected at this time point | 26.3 (27) | 41.4 (18) | 70.2 (19)

2. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Concentration (Tmax) of Dulaglutide
Description: Pharmacokinetic parameters were assessed on Day 1 in Part A and Days 1 and 22 in Part B.
Time Frame: Pre-dose and 12, 24, 48, 72, 96, 168, and 336 hours post-dose
Population: Participants in Part A and Part B who received at least 1 dose of study drug and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | 0.5 mg Dulaglutide (Part A-Healthy) | 0.75 mg Dulaglutide (Part A-Healthy) | 1.5 mg Dulaglutide (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM)
Number analyzed (Participants) | 10 | 11 | 11 | 11 | 11 | 10
hours
  Day 1 (Parts A and B) | 48.02 [12.02 to 48.02] | 48.00 [24.00 to 48.00] | 48.00 [24.00 to 48.00] | 48.00 [47.92 to 72.00] | 48.00 [24.00 to 72.00] | 71.98 [24.00 to 96.00]
  Day 22 (Part B only) | NA [NA to NA] — Part A participants did not have data collected at this time point | NA [NA to NA] — Part A participants did not have data collected at this time point | NA [NA to NA] — Part A participants did not have data collected at this time point | 48.00 [12.00 to 48.02] | 47.98 [24.00 to 48.00] | 48.00 [23.97 to 96.00]

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Time Zero to 336 Hours Postdose (AUC[0-336]) of Dulaglutide
Description: Pharmacokinetic parameters were assessed on Day 1 in Part A and Days 1 and 22 in Part B.
Time Frame: Pre-dose and 12, 24, 48, 72, 96, 168, and 336 hours post-dose
Population: Participants in Part A and Part B who received at least 1 dose of study drug and had evaluable AUC(0-336) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | 0.5 mg Dulaglutide (Part A-Healthy) | 0.75 mg Dulaglutide (Part A-Healthy) | 1.5 mg Dulaglutide (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM)
Number analyzed (Participants) | 10 | 11 | 11 | 11 | 11 | 10
nanograms*hours per milliliter (ng*h/mL)
  Day 1 (Parts A and B; n = 6, 10, 11, 3, 8, 4) | 4500 (42) | 6410 (14) | 11700 (12) | 3900 (7) | 5490 (19) | 10300 (16)
  Day 22 (Part B only; n = 6, 10, 10 | NA (NA) — Part A participants did not have data collected at this time point | NA (NA) — Part A participants did not have data collected at this time point | NA (NA) — Part A participants did not have data collected at this time point | 4720 (7) | 7030 (17) | 12500 (15)

4. Primary Outcome: Pharmacokinetics: Half-life of Dulaglutide
Description: Pharmacokinetic parameters were assessed on Day 1 in Part A and Days 1 and 22 in Part B.
Time Frame: Pre-dose and 12, 24, 48, 72, 96, 168, and 336 hours post-dose
Population: Participants in Part A and Part B who received at least 1 dose of study drug and had evaluable half-life data.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | 0.5 mg Dulaglutide (Part A-Healthy) | 0.75 mg Dulaglutide (Part A-Healthy) | 1.5 mg Dulaglutide (Part A-Healthy) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM)
Number analyzed (Participants) | 10 | 11 | 11 | 6 | 10 | 9
hours
  Day 1 (Parts A and B; n=6, 10, 11, 3, 8, 4) | 85.1 [50.8 to 244] | 84.5 [60.2 to 228] | 82.9 [63.8 to 104] | 122 [106 to 133] | 113 [63.9 to 222] | 88.5 [69.6 to 111]
  Day 22 (Part B only; n=NA, NA, NA, 6, 10, 9) | NA [NA to NA] — Part A participants did not have data collected at this time point | NA [NA to NA] — Part A participants did not have data collected at this time point | NA [NA to NA] — Part A participants did not have data collected at this time point | 97.6 [71.9 to 122] | 106 [70.4 to 139] | 105 [80.0 to 134]

5. Secondary Outcome: Part B - Pharmacodynamics: Area Under the Plasma Glucose Time Curve From Time Zero to 4 Hours Postmeal (gAUC[0-4])
Description: Pharmacodynamic parameters were assessed at baseline and on Days 3, 24, and 29 in Part B.
Time Frame: Baseline and Days 3, 24, and 29
Population: Participants in Part B who received at least 1 dose of study drug and had evaluable gAUC(0-4) data.
Measure: Mean (Standard Deviation); unit: millimoles*hours per liter (mmol*h/L)
Groups:
- Placebo (Part B-T2DM: Placebo administered to participants with T2DM once weekly SQ for 4 weeks in Part B
Arm/Group | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM) | Placebo (Part B-T2DM
Number analyzed (Participants) | 11 | 11 | 10 | 10
millimoles*hours per liter (mmol*h/L)
  Baseline | 44.3 (10.6) | 58.1 (11.7) | 53.4 (8.12) | 48.2 (7.00)
  Day 3 | 34.2 (6.19) | 41.2 (11.9) | 32.2 (4.87) | 46.1 (8.94)
  Day 24 | 34.7 (7.11) | 36.8 (7.08) | 30.5 (4.55) | 48.6 (9.10)
  Day 29 | 37.6 (9.11) | 38.1 (7.40) | 31.8 (4.57) | 46.9 (6.68)

ADVERSE EVENTS:
Groups:
- 0.5 mg Dulaglutide (Part A-Healthy): 0.5 milligrams (mg) dulaglutide administered once subcutaneously (SQ) to healthy participants in 1 of 3 treatment periods
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
- 0.75 mg Dulaglutide (Part A-Healthy): 0.75 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
- 1.5 mg Dulaglutide (Part A-Healthy): 1.5 mg dulaglutide administered once SQ to healthy participants in 1 of 3 treatment periods
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
- 0.5 mg Dulaglutide (Part B-T2DM): 0.5 mg dulaglutide administered to participants with Type 2 diabetes mellitus (T2DM) once weekly SQ for 4 weeks
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
- 0.75 mg Dulaglutide (Part B-T2DM): 0.75 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
- 1.5 mg Dulaglutide (Part B-T2DM): 1.5 mg dulaglutide administered to participants with T2DM once weekly SQ for 4 weeks
  Dulaglutide
  Placebo: Administered SQ in the placebo arms and to maintain the blind in the dulaglutide arms.
Arm/Group | Placebo (Part A-Healthy) | 0.5 mg Dulaglutide (Part A-Healthy) | 0.75 mg Dulaglutide (Part A-Healthy) | 1.5 mg Dulaglutide (Part A-Healthy) | Placebo (Part B-T2DM) | 0.5 mg Dulaglutide (Part B-T2DM) | 0.75 mg Dulaglutide (Part B-T2DM) | 1.5 mg Dulaglutide (Part B-T2DM)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/10 | 0/11 | 0/11 | 0/10 | 1/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/16 | 0/10 | 2/11 | 4/11 | 1/10 | 5/11 | 5/11 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A-Healthy) (N=16) | 0.5 mg Dulaglutide (Part A-Healthy) (N=10) | 0.75 mg Dulaglutide (Part A-Healthy) (N=11) | 1.5 mg Dulaglutide (Part A-Healthy) (N=11) | Placebo (Part B-T2DM) (N=10) | 0.5 mg Dulaglutide (Part B-T2DM) (N=11) | 0.75 mg Dulaglutide (Part B-T2DM) (N=11) | 1.5 mg Dulaglutide (Part B-T2DM) (N=10)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A-Healthy) (N=16) | 0.5 mg Dulaglutide (Part A-Healthy) (N=10) | 0.75 mg Dulaglutide (Part A-Healthy) (N=11) | 1.5 mg Dulaglutide (Part A-Healthy) (N=11) | Placebo (Part B-T2DM) (N=10) | 0.5 mg Dulaglutide (Part B-T2DM) (N=11) | 0.75 mg Dulaglutide (Part B-T2DM) (N=11) | 1.5 mg Dulaglutide (Part B-T2DM) (N=10)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days